CLINICAL TRIAL: NCT02591004
Title: Comparing Fetal Cerebral Blood Flow Between Magnesium Sulfate & Calcium Channel Blockers in Patients With Preterm Labor; a Randomized Controlled Trial.
Brief Title: Calcium Channel Blockers Compared to Magnesium Sulfate in Fetal Cerebral Blood Flow
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed M.Kamel, Lecturer of obstetrics & Gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A21102015
Record Dates: First submitted 2015-10-26; First posted 2015-10-29 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Preterm Labor; Cerebral Palsy
Keywords: Neuroprotection; calcium channel blockers; magnesium sulhate; Middle cerebral artery doppler
MeSH Terms: conditions — Obstetric Labor, Premature; Cerebral Palsy | interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magesium sulphate (Experimental): * Patients in group A will receive Magesium sulphate 4 gm intravenous (I.V) loading dose over 30 mins & 1 gm/ hour maintenance dose for 24 hours, or till labor occurs ( whichever occurs first).
  * Doppler on fetal middle cerebral artery
  Interventions: Drug: Magesium sulphate; Radiation: Doppler on fetal middle cerebral artery
- Nifedipine (Active Comparator): * Patients in group B will receive Nifedipine ( Epilat 10mg ® EIPICO Egypt ), as there is no recommended dose for the use of nifedipine as neuroprotectant, the dose given in this study will be same as that used for tocolysis. Nifedipine wil be given in a loading dose of 40 mg in the 1st hour (10mg will be given every 15 min), then a maintenance dose of 60mg /24 hours, divided in 3 doses.
  * Doppler on fetal middle cerebral artery
  Interventions: Drug: Nifedipine; Radiation: Doppler on fetal middle cerebral artery

INTERVENTIONS:
Drug: Magesium sulphate — *Experimental: Group A: Magesium sulphate 4 gm intravenous (I.V) loading dose over 30 mins & 1 gm/ hour maintenance dose for 24 hours, or till labor occurs ( whichever occurs first)
  Other Names: MgSo4
  Arms: Magesium sulphate
Drug: Nifedipine — *Active Comparator: Group B Nifedipine wil be given in a loading dose of 40 mg in the 1st hour (10mg will be given every 15 min), then a maintenance dose of 60mg /24 hours, divided in 3 doses
  Other Names: Epilat
  Arms: Nifedipine
Radiation: Doppler on fetal middle cerebral artery — both group A and group B: ultrasound doppler to measure the mean pulsility index (PI) and resistance index (PI) of the middle cerebral artery in the fetus twice, once before giving them the drug, and the other after 4 hours of starting the loading dose.

SUMMARY:
The aim of this study is to investigate the possible use of calcium channel as a neuroprotectant in cases with PTL. This will be done by comparing the effect they have on cerebral blood vessels with the already established MgSo4. They have been proven superior to magnesium sulphate in tocolysis, and they possess the mechanism of action that would allow for their theoretical use as neuroprotective agents.

DETAILED DESCRIPTION:
After internal review board approval from the obstetrics and gynecology department of Kasr Alainy hospital, 130 patients will be recruited in a randomized case control study. The patients will be recruited from the emergency admissions department, after fulfilling the recruitment criteria. In an independent case-control study the Sample size was calculated using an odds ratio of exposure to CP of 0.14 (95% CI 0.05-0.51) (Grether et.al, 1998), where the alpha level error was fixed at 0.5 and the power was set at 80%, the optimal sample size was calculated to be 65 patients in each arm.

Patients will be randomized on admission by nurse in labor ward into either one of two groups. Group A will receive MgSo4, while group B will receive Nifedipine ( Epilat 20mg ® EIPICO Egypt ). Randomization will be achieved through a computer generated randomization table. Recruitment will continue till 65 patients will be allocated to each group.

Patients in group A will receive 4 gm intravenous (I.V) MgSo4 loading dose over 30 mins & 1 gm/ hour maintenance dose for 24 hours, or till labor occurs ( whichever occurs first) , this does is given in accordance with Australian Research Centre for Health of Women and Babies, 2010, for using MgSo4 for neuroprotection against CP.

While patients in group B will receive Nifedipine ( Epilat 10mg ® EIPICO Egypt ), as there is no recommended dose for the use of nifedipine as neuroprotectant, the dose given in this study will be same as that used for tocolysis. Nifedipine wil be given in a loading dose of 40 mg in the 1st hour (10mg will be given every 15 min), then a maintenance dose of 60mg /24 hours, divided in 3 doses (Hösli et.al, 2014).

The ability of the MgSo4 as a neuro protectant is dependent on its cerebral vasodilating effects (Magee et.al,2011; Macdonald et.al, 2004), therefore we propose to measure the mean pulsility index (PI) and resistance index (PI) of the middle cerebral artery in the fetus twice, once before giving them the drug, and the other after 4 hours of starting the loading dose. All ultrasound and power doppler examinations will be carried out by the same investigator, using the Voluson 730 machine (GE Healthcare Austria GmbH, Seoul, Korea). Sample size calculation was done using Stats Direct statistical software version 2.7.2 for MS Windows, StatsDirect Ltd., Cheshire, UK.

ELIGIBILITY:
* Inclusion Criteria:

  * in imminent preterm labour ( , >4cm dilated, cervical effacement > 60%).
  * < 32 weeks gestational age.
* Exclusion Criteria:

  * patients will be excluded from the study if the gestational age was > 32 weeks
  * intrauterine fetal death
  * multiple gestation
  * fetal malformations where only palliative care is needed
  * placental abruption
  * Chorioamnionitis
  * pre-ecplamsia, or diabetes
  * suspected fetal compromise diagnosed by ultrasound or CTG requiring delivery, -any indication for caesarean section
  * fetal growth restriction
  * Also any contraindication to the use of Nifedipine e.g maternal cardiac disease, allergy to Nifedipine, hypotension, or hepatic dysfunction
  * Contraindications To MgSo4 use as Myasthenia Gravis, progressive muscle weakness ,allergy to MgSo4, severe renal impairment & heart block.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2015-12; Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
difference in mean doppler indicies of middle cerebral artery of fetus between both groups | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Kamel, M.D., Principal Investigator — Lecturer of obstetrics & Gynecology; Wafaa Eldesouky, M.D., Principal Investigator — Lecturer of obstetrics & Gynecology
Locations (1):
- 11562, Cairo, Egypt

REFERENCES:
- [Background] Magee L, Sawchuck D, Synnes A, von Dadelszen P; MAGNESIUM SULPHATE FOR FETAL NEUROPROTECTION CONSENSUS COMMITTEE; MATERNAL FETAL MEDICINE COMMITTEE. SOGC Clinical Practice Guideline. Magnesium sulphate for fetal neuroprotection. J Obstet Gynaecol Can. 2011 May;33(5):516-529. doi: 10.1016/S1701-2163(16)34886-1. PMID 21639972
- [Background] Hosli I, Sperschneider C, Drack G, Zimmermann R, Surbek D, Irion O; Swiss Society of Obstetrics and Gynecology. Tocolysis for preterm labor: expert opinion. Arch Gynecol Obstet. 2014 Apr;289(4):903-9. doi: 10.1007/s00404-013-3137-9. Epub 2014 Jan 3. PMID 24385286
- [Background] Australian Research Centre for Health of Women and Babies. Antenatal Magnesium Sulphate Prior to Preterm Birth for Neuroprotection of the Fetus, Infant and Child - National Clinical Practice Guidelines. Adelaide. ARCH; 2010 [www.adelaide.edu.au/arch/].
- [Background] Macdonald RL, Curry DJ, Aihara Y, Zhang ZD, Jahromi BS, Yassari R. Magnesium and experimental vasospasm. J Neurosurg. 2004 Jan;100(1):106-10. doi: 10.3171/jns.2004.100.1.0106. PMID 14743919
- [Background] Grether J, Hirtz D, McNellis D, Nelson K, Rouse DJ. Tocolytic magnesium sulphate and paediatric mortality. Lancet. 1998 Jan 24;351(9098):292; author reply 293. doi: 10.1016/S0140-6736(05)78239-8. No abstract available. PMID 9457123